CLINICAL TRIAL: NCT07238907
Title: A Multi-center Retrospective Study of Inotuzumab Ozogamicin Treating Acute B-cell Lymphoblastic Leukemia
Brief Title: A Multi-center Retrospective Study of INO Treating B-ALL
Status: Active, not recruiting | Type: Observational
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Jin Wang, chief physician, MD, PhD, Ruijin Hospital
Other Study IDs: RJ-ALL 2025-B03
Record Dates: First submitted 2025-09-22; First posted 2025-11-20 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Acute Lymphoblastic Leukaemia; Acute Lymphoblastic Leukaemias (ALL); Inotuzumab Ozogamicin; Venetoclax
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Inotuzumab Ozogamicin

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- observation group
  Interventions: Drug: Inotuzumab Ozogamicin

INTERVENTIONS:
Drug: Inotuzumab Ozogamicin — All patients have received Inotuzumab Ozogamicin

SUMMARY:
This multi-center retrospective study aims to evaluate the efficacy and safety of inotuzumab ozogamicin in adults B-ALL of different subgroups. This study is a retrospective study. Data will be collected from Electronic Medical Record, interventions will not be implemented on patients.

ELIGIBILITY:
Inclusion Criteria:

* Age between ≥16 and ≤80 years at screening, no gender restrictions
* Be diagnosed with B-ALL
* Appropirate organ function, meeting the following criteria:

  1. Aspartate aminotransferase (AST) ≤3 times the upper limit of normal (ULN);
  2. Alanine aminotransferase (ALT) ≤3 times ULN;
  3. Total bilirubin ≤2 times ULN (for patients with Gilbert's syndrome, total bilirubin ≤3.0 times ULN and direct bilirubin ≤1.5 times ULN);
  4. Serum creatinine ≤1.5 times ULN, or creatinine clearance ≥60 mL/min (using the Cockcroft-Gault formula);
  5. Left ventricular ejection fraction (LVEF) ≥50%;

Exclusion Criteria:

* Active infection at screening.
* Any of the following cardiac conditions:

  1. NYHA Class III or IV congestive heart failure;
  2. Severe arrhythmia requiring treatment;
  3. Uncontrolled hypertension or pulmonary hypertension despite standard therapy;
  4. Unstable angina;
  5. Myocardial infarction, bypass surgery, or stent placement within six months before cell retransfusion;
  6. Clinically significant valvular disease;
  7. Other cardiac conditions deemed unsuitable by the investigator;
* History of epilepsy, cerebellar disease, or other active central nervous system disorders;
* History of hypersensitivity to any component of the investigational product.
* Life expectancy of less than three months;
* Other conditions deemed unsuitable for participation in this clinical trial by the investigator.

Ages: 16 Years to 80 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patients received INO-based therapy in all participant center of this study
Sampling Method: Non-Probability Sample
Enrollment: 102 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
overall response rate | Till the end of the study, up to 12 months
  The proportion of patients who reach CR/CRi.Bone marrow of every patient will be analysed by multiparameter flow cytometry or/and RT-qPCR for MRD evaluation.

SECONDARY OUTCOMES:
minimal residual disease negativity rate | Till the end of the study, up to 12 months
  The proportion of patients who reach MRD negative in all patients reached CR/CRi.Bone marrow of every patient will be analysed by multiparameter flow cytometry or/and RT-qPCR for MRD evaluation.
overall survival | Till the end of the study, up to 12 months
  Interval from the date of the feedback to the time of death due to any reason. Evaluation of OS will be based on follow-up results.
Relapse-free survival | Till the end of the study, up to 12 months
  Interval from the date of reception of the INO-based therapy to the time of hematological recurrence or death from any cause. Evaluation of RFS will be based on follow-up results.
Hematological toxicity: neutropenia, thrombocytopenia, febrile neutropenia, anemia, bone marrow suppression Non hematological toxicity: SOS,TLS, peripheral edema, fever, fatigue, MODS, infection, liver dysfunction, renal dysfunction et al. | Till the end of the study, up to 12 months
  Hematological toxicity includes: neutropenia, thrombocytopenia, febrile neutropenia, anemia, and bone marrow suppression Non hematological toxicity includes sinus obstruction syndrome(SOS), tumor lysis syndrome(TLS), peripheral edema, fever, fatigue, multiple organ dysfunction syndrome(MODS), infection, liver dysfunction, renal dysfunction, abnormal blood electrolytes, and infusion reactions.
  All AEs will be assessed by CTCAE v5.0

CONTACTS AND LOCATIONS:
Locations (1):
- Ruijin Hospital, Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided